CLINICAL TRIAL: NCT00278824
Title: A Double-Blind, Placebo-Controlled, Proof-of-Concept Study to Evaluate the Efficacy of CHADD™ Applied Over a Transdermal Fentanyl Patch for the Treatment of Breakthrough Pain in Patients With Moderate to Severe Non-malignant Chronic Pain
Brief Title: Fentanyl Transdermal Patch With CHADD™ for Breakthrough Pain in Patients With Moderate to Severe Non-Malignant Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty identifying and enrolling eligible patients
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZCM-201
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Pain
Keywords: Chronic Pain; Pain
MeSH Terms: conditions — Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 50 mcg/hr matrix fentanyl patch (Experimental): active 50 mcg/hr ZR-02-01 matrix transdermal fentanyl patch (20 cm2)
  Interventions: Drug: Matrix Transdermal Fentanyl/CHADD Drug Delivery System
- Placebo Patch (Placebo Comparator): placebo (20 cm2) will be indistinguishable in size, shape, and appearance to the active matrix fentanyl patch
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: Matrix Transdermal Fentanyl/CHADD Drug Delivery System — Patch applied every 3 days for 15 days
  Other Names: ZR-02-01; Fentanyl Transdermal Matrix Patch
  Arms: 50 mcg/hr matrix fentanyl patch
Drug: Placebo Patch — Placebo patch applied every 3 days for 15 days
  Other Names: Placebo Matrix Patch
  Arms: Placebo Patch

SUMMARY:
A multi-center study to evaluate the efficacy of CHADD (Controlled Heat-Assisted Drug Delivery) applied over a 50 mcg/hr ZR-02-01 matrix transdermal fentanyl patch for the treatment of breakthrough pain in adult patients with moderate to severe non-malignant chronic pain. The open-label study arm will last up to 12 days. The double-blind arm will last up to 15 days. Eligible patients who complete the open-label arm will be allowed to enroll in the double-blind study arm.

DETAILED DESCRIPTION:
ZARS Pharma is developing a Matrix Transdermal Fentanyl/CHADD (Controlled Heat-Assisted Drug Delivery) Drug Delivery System to be used for the treatment of chronic and breakthrough pain. The Matrix Transdermal Fentanyl/CHADD Drug Delivery System has been designed to provide long-term delivery of fentanyl for the treatment of chronic pain as well as intermittent increases in fentanyl concentrations for the treatment of breakthrough pain. Breakthrough pain is defined as a transitory exacerbation of pain that occurs on a background of otherwise stable pain in a patient receiving chronic opioid therapy.

Matrix Transdermal Fentanyl/CHADD Drug Delivery System has 2 components: a matrix transdermal fentanyl patch (the ZR-02-01 patch in doses of 25, 50, 75 and 100 mcg/hr) with corresponding thin film dressing (ie, overlay) and the CHADD (Controlled Heat-Assisted Drug Delivery).

The matrix transdermal fentanyl patch provides a continuous delivery of fentanyl over 72 hours, in a manner similar to Duragesic®. During a breakthrough pain episode, a CHADD unit is placed over (adhered to) the matrix transdermal fentanyl patch. The CHADD is a thin patch-like chemical heating device that generates a controlled level of heat for approximately 15-20 minutes. The application of heat delivers increased amounts of fentanyl when applied over the ZR-02-01 matrix transdermal fentanyl patch.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 through 70 years of age.
* Patient has moderate to severe non-malignant chronic pain.
* Patient is opioid-tolerant, requires treatment with chronic opioids and is currently taking a dose of 50 mcg/hr transdermal fentanyl for the treatment of chronic pain. Patient must have been taking this dose for at least 2 weeks.
* Patient must be experiencing 1 to 4 episodes of target breakthrough pain (breakthrough pain that is related to the patient's chronic pain condition) a day while taking a dose of 50 mcg/hr transdermal fentanyl.

Exclusion Criteria:

* Patient has active cancer.
* Patient has a history of substance abuse or has a substance abuse disorder.
* Patient is pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2006-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Patient's rating of pain intensity (NRS), the patient's evaluation of pain relief using a 5-point verbal rating scale (VRS), and the patient's global satisfaction assessment. | 0, 15, 20, 60 minutes
  Efficacy will be evaluated by the patient's rating of pain intensity using an 11-point numerical rating scale (NRS), the patient's evaluation of pain relief using a 5-point verbal rating scale (VRS), and the patient's global satisfaction assessment.

SECONDARY OUTCOMES:
Adhesion assessment | 3 days
  An adhesion assessment will be conducted by the patient at each CHADD removal.
Pain Relief | 15, 30, 60 minutes
  Patient's evaluation of pain relief using a 5-point verbal rating scale (VRS)
Patient's Global Satisfaction Assessment | 60 minutes
  Patients completed a global satisfaction assessment 60 minutes after CHADD application. Patients were asked to assess their overall satisfaction with the CHADD throughout the 60 minute application period for the treatment of their breakthrough pain using the following 5-point scale: 0=not satisfied,
  1=somewhat satisfied, 2=moderately satisfied, 3=very satisfied, and 4=completely satisfied.
Number of participants with adverse events | 15 days
  The frequency of adverse events, severity, and relationship to study drug was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn R Webster, MD, Principal Investigator — Lifetree Clinical Research
Locations (15):
- United States (15):
  - Arizona Reserach Center, Phoenix, Arizona
  - Florida's Institute of Clinical Research, Jacksonville, Florida
  - Drug Studies America, Marietta, Georgia
  - Pain & Rehabilitation Clinic of Chicago, Chicago, Illinois
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Medical Advanced Pain Specialists, Minneapolis, Minnesota
  - Pain Management Associates, Independence, Missouri
  - Analgesic Development Ltd., New York, New York
  - Southeast Research Institute, Charlotte, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Pain Consultants of Oregon, PC, Eugene, Oregon
  - Allegheny Pain Management, Altoona, Pennsylvania
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Advanced Pain Management, Virginia Beach, Virginia